CLINICAL TRIAL: NCT05382962
Title: iCanCope With Post-Operative Pain (iCanCope PostOp): Development of a Smartphone-based Pain Self-management Program for Adolescents Following Surgery
Brief Title: iCanCope With Post-Operative Pain (iCanCope PostOp)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinician Scientist, Clinical Nurse Specialist/NP, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1000070021
Record Dates: First submitted 2022-05-11; First posted 2022-05-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Pain, Chronic; Pain, Chronic Post-Surgical
Keywords: paediatric chronic pain; post-surgical
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomization will be done independently at each site (i.e., SickKids and Boston Children's Hospital), and will be stratified by type of surgery (i.e. pectus repair, scoliosis). Following consent and measure completion, study staff will randomize the participant using a 1:1 randomization allocation to intervention vs. control groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: iCanCope Post-Op App (Experimental): Adolescents randomized to the intervention group will receive the iCanCope PostOp app, in addition to usual care. Both groups will complete measures at pre-operative appointments following consent and randomization (6-8 weeks prior to surgery, T0), at 1-week pre-op (T1), 2-week post-op, (T2) and 4-week post-op (T3), and 12-week post-op (T4).
  Interventions: Behavioral: iCanCope Post Op Application
- Control: Usual Care (No Intervention): Adolescents randomized to the control group will receive usual care. Both groups will complete measures at pre-operative appointments following consent and randomization (6-8 weeks prior to surgery, T0), at 1-week pre-op (T1), 2-week post-op, (T2) and 4-week post-op (T3), and 12-week post-op (T4).

INTERVENTIONS:
Behavioral: iCanCope Post Op Application — The iCanCope program is designed to enhance pain self-management and self-efficacy, defined as perception of one's ability to successfully produce a desired effect in a task or behavior affecting their life. The intervention will be delivered on the iOS or Android smartphone platform depending on the participant's device. Usage of app features will be centrally tracked by the research team using Analytics Platform to Evaluate Effective Engagement (APEEE), developed at the Centre for Global eHealth Innovation. Participants will receive alerts through iCanCope to complete a pain diary check-in once per week preoperatively, twice per day over the initial 2-week postoperative period, and once per day for the subsequent 2-week period.
  Arms: Intervention: iCanCope Post-Op App

SUMMARY:
There are few applications available in the community to help teenagers manage pain after surgery. The focus of this study is to better understand the pain experience of children after having surgery and to design a Smartphone app called "iCanCope with Post-Operative Pain" (iCanCope PostOp), to help children and parents to better manage pain at home after surgery. The app will help keep track of pain, provide information about the teenager's surgery and provides "in-the-moment" advice wherever and whenever the patient needs it.

DETAILED DESCRIPTION:
More than 80,000 Canadian children undergo surgery each year. Despite evidence-based pain management and clinical standards, moderate to severe postoperative pain in children is common. Inadequate postoperative pain management contributes to poor health outcomes, increased opioid use, and the development of chronic postsurgical pain. Successful postoperative pain management requires regular monitoring and treatment of pain after hospital discharge. Smartphones are nearly ubiquitous, and growing evidence supports their use to overcome barriers to pain care. Computerized clinical decision support systems (CDSS) can improve pain self-management by tracking symptoms over time and offering tailored evidence-informed pain management advice based on standardized algorithms. A comprehensive and sustainable approach is needed to address poorly managed pediatric postoperative pain in the home setting. To address these gaps in care, we are developing "iCanCope with Post-Operative Pain" (or iCanCope PostOp), a smartphone-based CDSS app that provides remote, in-the-moment advice to improve pain and health-related quality of life (HRQL) for adolescents following surgery.

ELIGIBILITY:
Inclusion Criteria:

1. aged 12 to 18 years;
2. own a smartphone compatible with the iCanCope app (iOS or Android);
3. diagnosed with adolescent idiopathic scoliosis or pectus carinatum or pectus excavatum;
4. are able to speak and read English; and
5. scheduled to undergo scoliosis or minimally invasive pectus repair surgery.

Exclusion Criteria:

1. significant cognitive impairment or other co-existing medical condition that could limit the ability to use the iCanCope app, as identified by their health care provider;
2. participated in a previous study of iCanCope PostOp;
3. a diagnosed chronic pain condition not related to the surgical condition; or

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Participant Accrual and Dropout Rates | 12 weeks
  This will be centrally tracked by the clinical research project coordinator (CRPC).
Intervention fidelity | 12 weeks
  Any issues or difficulties encountered during implementation of the intervention, control strategy, or outcome measures will be tracked throughout the study by the CRPC.
Acceptability and Satisfaction | 12 weeks
  Participants in the intervention arm will complete the Acceptability e-scale (AES) post-intervention. In addition, a subset of participants from the intervention group will be offered to participate in a qualitative feedback interview to further explore acceptability and satisfaction of the intervention.
Engagement with Intervention | 12 weeks
  Google Analytics will track patterns of app and website usage.

SECONDARY OUTCOMES:
Pain intensity and interference | 12 weeks
  Measured using the short form Brief Pain Inventory (BPI), a 15-item tool that measures pain intensity and impact on functioning.
Sleep Functioning | 12 weeks
  Measured with the PROMIS Pediatric Sleep Disturbance - Short Form 4a, a 4-item measure for assessing sleep disturbance. Each item asks the child receiving care to rate the severity of his or her sleep disturbance during the past 7 days. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Physical Function | 12 weeks
  Measured using the PROMIS Pediatric Mobility SF, an 8-item questionnaire designed to investigate the general impact that the patient's lower limbs mobility had on their daily activity tasks (such as playing with friends or walking up the stairs). Each item is scored from 1 (not able to do it0 to 5 (with no trouble). As per PROMIS guidelines, raw score is calculated as the sum of each item score. Scale score was calculated from raw score using the PROMIS conversion table.
Depressive Symptoms | 12 weeks
  Measured using the PROMIS Pediatric Depressive Symptoms SF, an 8-item questionnaire designed to determine how often one is experiencing specific depressive symptoms in the past 7 days. Each item on the measure is rated on a 5-point scale (1=never; 2=almost never; 3=sometimes; 4=often; and 5=almost always) with a range in score from 14 to 70 with higher scores indicating greater severity of depression.
Anxiety | 12 weeks
  Measured using the PROMIS Anxiety SF, the 13-item questionnaire that assesses the pure domain of anxiety in children and adolescents. Each item asks the child receiving care to rate the severity of his or her anxiety during the past 7 days. Each item on the measure is rated on a 5-point scale (1=never; 2=almost never; 3=sometimes; 4=often; and 5=almost always) with a range in score from 13 to 65 with higher scores indicating greater severity of anxiety.
Overall health | 12 weeks
  Measured using the Patients Global Impression of Change (PGIC), that reflects a patient's belief about the efficacy of treatment. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
School attendance | 12 weeks
  Self-report, investigator developed

OTHER OUTCOMES:
Medication utilization | 12 weeks
  Self-report, investigator developed (Prescribed and over-the-counter pain medication)
Health care utilization | 12 weeks
  Self-report, investigator developed (Health care visits to various providers, Hospital stay, prescriptions, and admission data from EMR)
Child Surgical Worries | 2 weeks
  Measured using the Child Surgical Worries Questionnaire, a 27-item self-report measure assessing worries caused by hospitalization and surgery. Patients rate how worried they are about various situations, using the following scale: 0=not at all worried, 1=a little worried, 2=moderately worried, 3=considerably worried, 4=extremely worried.
Parent Catastrophizing (Parent Outcome) | 12 weeks
  Measured using the Pain Catastrophizing Scale - Parent (PCS-P), a 13-item questionnaire concerning the different thoughts and feelings parents may have when their child experiences pain. Items assessing catastrophic thoughts and feelings about their child's pain use a Likert-type 5-point scale (0 = "not at all" to 4 = "extremely"). The PCS-P yields three subscale scores for rumination, magnification, and helplessness, as well as a total score ranging from 0 to 52.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stinson, RN, PhD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Boston Children's Hospital, Boston, Massachusetts, United States
- Hospital for Sick Children, Toronto, Ontario, Canada